CLINICAL TRIAL: NCT00933556
Title: A Pilot Randomized Trial to Determine the Efficacy of a Probiotic, VSL#3 for Reducing Colonization by Vancomycin-resistant Enterococcus (VRE)
Brief Title: A Pilot Trial to Determine the Efficacy of VSL#3 for Reducing Colonization by VRE
Acronym: PROVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-2008-0023
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Anti-biotic Resistance
Keywords: infection; probiotics
MeSH Terms: conditions — Infections | interventions — Sugars; trichlorosucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- probiotic (Experimental): subjects will be given a powder formulation of a probiotic VSL#3 to be taken once a day, at a dose of 6 gms
  Interventions: Dietary Supplement: VSL#3
- sugar pill (Placebo Comparator): placebo identical to the active product will be given
  Interventions: Dietary Supplement: sugar pill (placebo)

INTERVENTIONS:
Dietary Supplement: VSL#3 — 6 gms of powder formulation to be given once a day for 4 weeks
  Other Names: yoplait; activia
  Arms: probiotic
Dietary Supplement: sugar pill (placebo) — placebo identical to the active product will be given
  Other Names: splenda
  Arms: sugar pill

SUMMARY:
The purpose of this study is to investigate the feasibility, safety and efficacy of oral probiotic, VSL#3 versus oral placebo for reducing colonization by VRE.

DETAILED DESCRIPTION:
Healthcare-associated infections are an important threat to patient safety. Currently, between 5 and 10 percent of patients admitted to acute care hospitals acquire one or more infections; healthcare-associated infections affect approximately 2 million patients each year in the United States, result in 90,000 deaths, and are associated with an added cost of $4.5 to $5.7 billion per year. Seventy percent of healthcare-associated infections are caused by antimicrobial resistant bacteria, such as vancomycin-resistant enterococcus (VRE), resulting in increased antimicrobial usage, morbidity and mortality, making prevention of multiresistant bacteria essential.

Eradication of colonization has been shown to greatly reduce infection; however, there are no reliable means of providing sustained eradication of colonization. No effective means of eradicating VRE intestinal colonization exist.

Probiotics containing strains of lactobacilli represent a novel approach to the prevention and control of antimicrobial resistance and have been studied extensively for a variety of infections. Even though various studies have shown probiotics to be effective for prevention of vaginal infections, urinary tract infections, etc no studies have examined the potential of probiotics to eradicate colonization by resistant pathogens, such as VRE.

ELIGIBILITY:
Inclusion Criteria:

* subjects will be male or female
* 18 years of age or older
* may or may not be hospitalized
* able to take oral medications
* have been found to be colonized with VRE or at high risk of being colonized by VRE and are not taking antibiotics

Exclusion Criteria:

* people on antibiotics will not be eligible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The main outcomes will be the proportion of patients colonized with VRE at 4 weeks, 8 weeks, 12 weeks and 24 weeks following start of treatment. | 24 weeks

SECONDARY OUTCOMES:
Incidence of clinical infections will be assessed in the one year following enrollment into the study. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nasia Safdar, MD, MS, Principal Investigator — University of Wisconsin Department of Medicine (Infectious Disease)
Locations (1):
- University of wisconsin hospital, Madison, Wisconsin, United States